CLINICAL TRIAL: NCT07085845
Title: Self-Sampling to Optimize Anal Lesion Outcomes (SOLO) Pilot
Brief Title: The Self-Sampling Pilot Study
Acronym: SOLOPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Alan Nyitray, PhD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PRO00055613
Record Dates: First submitted 2025-07-10; First posted 2025-07-25 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Anus
Keywords: squamous cell carcinoma of the anus; self-sampling; swab performance characteristics
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Individuals in the intervention arm will self-sample with a swab and insert the swab 5 cm into the anus.
  Interventions: Other: Inserting a swab 5 cm into the anus during self-sampling
- Control arm (Active Comparator): Individuals in the control arm will self-sample with a swab and insert the swab 3 cm into the anus.
  Interventions: Other: Self-sampling with a swab by inserting the swab 3 cm into the anus.

INTERVENTIONS:
Other: Inserting a swab 5 cm into the anus during self-sampling — The swab will be inserted into the anus by the lay individual. The individual will insert the swab to a depth of 5 cm to collect anal exfoliated cells.
  Arms: Intervention arm
Other: Self-sampling with a swab by inserting the swab 3 cm into the anus. — The swab will be inserted into the anus by the lay individual. The individual will insert the swab to a depth of 3 cm to collect anal exfoliated cells.
  Arms: Control arm

SUMMARY:
The investigators will test the cytological performance of a nylon-flocked swab at two insertion depths in the anus, 3 cm and 5 cm, to determine which insertion depth is better at collecting cells from the squamocolumnar junction (SCJ), an anatomic site that is particularly vulnerable to carcinogenic transformation. The investigators hypothesize that the 5 cm insertion will result in a higher quality specimen with cells from the SCJ. However, the deeper swab insertion may affect end user acceptability without increasing adequacy or quality.

DETAILED DESCRIPTION:
An important component of our parent SOLO study is the testing of two different kinds of swabs, nylon-flocked and Dacron, for cytological adequacy and end user acceptability within a self-sampling and clinician-sampling context. The investigators chose a nylon-flocked (NF) swab given its high adequacy in our prior study; however, this NF swab is unlikely to be available for clinical use in the future due to recent changes in the manufacturer's priorities. Since the parent study results need to be widely generalizable and relevant to anal cancer screening, The investigators need to use a different NF swab model and assess its cytological performance characteristics in a pilot study before beginning the parent study.

Given our prior success with a NF swab developed by Copan Italia s.p.a. (Brescia, Italy) the investigators will test the feasibility of a new Copan swab developed for anal cancer screening. The investigators will test the cytological performance of the swab at two insertion depths, 3 cm and 5 cm, to determine which insertion depth is better at collecting cells from the squamocolumnar junction (SCJ), an anatomic site that is particularly vulnerable to carcinogenic transformation. The investigators hypothesize that the 5 cm insertion will result in a higher quality specimen with cells from the SCJ. However, the deeper swab insertion may affect end user acceptability without increasing adequacy or quality.

The investigators will test the new swab with 60 individuals who were participants in a prior study and who agreed to be contacted for follow-up studies. Individuals will be randomized to use the new NF swab with either a 3 cm or 5 cm insertion depth. After consenting, individuals will receive written instructions and then conduct the self-sampling in private. Staff will take the swab in PreservCyt® to the Medical College of Wisconsin Tissue Bank where it will be aliquoted for assessment of cytology and reflex human papillomavirus (HPV) testing at Wisconsin Diagnostic Labs.

The investigators have one objective: To ensure the use of a swab in SOLO that is comparable to the originally proposed swab for SOLO, determine the preliminary performance characteristics of the new NF swab. • H1: A higher proportion of the new NF swabs with 5 cm insertion will have SCJ cells compared to the NF swab for 3 cm insertion.• H2: A higher proportion of the new NF swabs with 5 cm insertion will be adequate for cytopathology interpretation compared to the NF swab for 3 cm insertion.• H3: The new NF swab will have acceptability/pain performance commensurate with the originally proposed NF swab and the 5 cm insertion depth will have similar acceptability/pain performance as the 3 cm insertion depth. Our expected outcomes are cytological preliminary performance characteristics of the new NF swab in addition to user acceptability. These outcomes will help ensure the use of a viable swab in the parent study that is relevant in future anal cancer screening programs.

Recruitment Potential participants will be recruited first from the group of individuals who consented into the prior Prevent Anal Cancer (PAC) Self-Swab Study (PRO00032999) and then indicated an interest in a follow-up study (n=126). The investigators will enroll those aged ≥ 35 years. If the initial recruitment results in fewer than 60 people, the investigators will recruit by placing print materials in local gay-friendly businesses. The material will mention the study is recruiting for an anal cancer screening study. Recruitment material will be approved by a Medical College of Wisconsin (MCW) Institutional Review Board (IRB). The SOLO Study Coordinator in Milwaukee will oversee recruitment activity. The investigators will record recruitment activities.

Consenting Potential participants will be screened using an online computer-assisted self-interview (CASI). Those who are eligible will be asked to leave contact information. Study staff will contact eligible individuals, provide an overview of the pilot study, and invite the individual to a schedule a consenting session which will be followed by the cytology screening at the Curative Building on the MCW campus. Those who are not eligible will be thanked for their interest and provided links to vetted anal cancer education websites. Minimal Protected Health Information (PHI) will be collected in the eligibility survey.

At the consenting session staff will first ask the eligible individual to confirm their email address, name, and birthdate. The session will occur in a closed office and include information about 1) high rates of anal cancer in some populations, 2) anal cancer screening and the role of swabbing, 3) pilot study activities, and 4) the potential harms and benefits of participation. The staff member obtaining consent will emphasize that participation is voluntary and that participants can choose to join and, if desired, leave the pilot study at any point without any repercussions. Prior to obtaining their signature, the staff member will ask the individual if they have any questions and, if not, to briefly review their understanding of their participation by asking simple questions about the pilot study to be sure the information was clearly understood.

Individuals agreeing to provide consent will sign an informed consent form (ICF) hard copy. It will be photocopied with the copy given to the participant.

Study Design This pilot feasibility study will use a randomized controlled trial design. Randomization Consented individuals will be randomized to either the intervention (5 cm insertion depth) or the control (3 cm insertion depth) arm using a number generator in REDCap. If the number is .0000 to .4999, the individual will be assigned to the intervention condition. If the number is .5000 to .9999, the individual will be assigned to the control condition. The participant is considered enrolled in the pilot study when they sign a consent form and are randomized to either the intervention or control arm.

Cytology Sampling The cytology sampling will occur immediately after randomization. In preparation, staff will have created two cytology collection kits (labeled as Kit A or Kit B) each containing swabbing instructions, a swab, ThinPrep vial, and gloves. Kit A and Kit B will have identical contents except that Kit A will have a swab with a mark 5 cm from the swab tip and Kit B will have a swab with a mark 3 cm from the swab tip. Clinical staff will review the sampling instructions with the individual and then show them to a bathroom in the Curative Building on the MCW campus with a locking door where the individual will do the self-sampling with sampling instructions available. Individuals will be instructed to take the cap off the vial, put on gloves, remove the swab from the packaging, hold the swab at the mark on the shaft of the swab (which corresponds to either 3 cm or 5 cm), get in a comfortable position, insert the swab gently all the way to the mark, begin to twirl the swab clockwise and counterclockwise, and apply pressure to the anal canal walls, while removing the swab as they count slowly to 10.After swabbing, the participant will put the swab in 20 mL of PreservCyt® solution, agitate and twirl it in the solution for 10 seconds, and then remove the swab while pressing against the sides of the vial. The swab will be discarded, the vial cap replaced, and the vial inserted back into the kit and returned to the staff member. Participants will be instructed to wash their hands.

Participants will complete a short CASI in the consenting office in private on their phone (or hard copy if they prefer) immediately after their self-sampling to assess the swabbing experience, including discomfort and pain, using validated questions. Clinic staff will assist individuals with technology limitations. For those who do not show up for their consenting and cytology appointment, a member of the study team will contact them twice to reschedule within 2 months of their original appointment date.

Kit Processing, Cytopathology, and Reflex HPV Testing Staff will walk the cytology kit to the MCW Tissue Bank who will process the PreservCyt liquid by removing a 0.5 mL aliquot. The remaining specimen will be kept in the original vial for cytopathology.

The remaining specimen will be delivered to Wisconsin Diagnostic Labs (Milwaukee, Wisconsin) which uses the COBAS 4800 system for cytology reading. Cytology findings will use the Bethesda System with classification as follows: negative for intraepithelial lesions; atypical squamous cells of undetermined significance (ASCUS) or atypical squamous cells, cannot rule out high-grade squamous intraepithelial lesion; low-grade squamous intraepithelial lesion; or high-grade squamous intraepithelial lesion. Reflex HPV testing will be conducted for all abnormal (i.e., ≥ ASCUS) specimens.

Anal cytology is approved for use in anal cancer screening. Thus, individuals will be given the cytopathology results and any HPV reflex testing results through the individual's preferred mode of communication; however, regardless of the result, all individuals will be encouraged to seek medical advice about their results. Currently, there is no FDA approval for anal self-sampling, thus, the cytology results should not be used to guide care or referrals.

End of Pilot Study Definition An individual is considered to have completed the study if they have completed the post-cytology survey. Those who participated in the pilot study will not be eligible or involved in the parent SOLO study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 35 years.
2. Must be either:

   1. A sexual minority man, or
   2. A woman who has a different identity than the sex she was born with.
3. Resides in the Milwaukee metropolitan area.
4. Speak and understand English.
5. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Presence of any contraindicating severe anal disease or condition, e.g., anal stenosis.

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nyitray, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Curative Building, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
This Self-sampling to Optimize anal Lesion Outcomes (SOLO) pilot study will produce quantitative data generated from surveys with 60 participants. We will also collect data on intervention performance, biospecimen collection, and laboratory assays. Data from the 60 persons will be collected at 1 time point, the cytology appointment.
  To protect research participant identities, only de-identified individual quantitative data will be made available for sharing.
  The final datasets will include quantitative data as delineated in 1.A. We will share de-identified individual participant-level data. We will use typical strategies such as "safe harbor" methods that remove all protected health information (e.g., name, address, and contact information) per MCW policy AD.HP.090. Informed consent forms will reflect those plans. In circumstances where small sample sizes may allow identification of research participants, only summarized data will be made available for sharing.
Supporting Information: Study Protocol, ICF
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication. The duration of preservation and sharing of the data will be a minimum of 10 years.
Access Criteria: The openICPSR provides metadata, persistent identifiers using ICPSR ID numbers and DOI, and long-term access. The repository is supported by the Inter-university Consortium for Political and Social Research (ICPSR) and datasets are available under a Creative Commons Attribution 4.0 International (CC BY 4.0) License. The dataset will be discoverable online by anyone through a standard web search of the study-level metadata as well as the persistent pointer from the ICPSR ID and DOI to the dataset.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (10.4) | 56.1 (11.6) | 55.3 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 23 | 26 | 49
  Trans Man | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 19 | 22 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Presence of Squamocolumnar Cells
Description: The presence of cells from the squamocolumnar junction will be assessed in each specimen (Yes/No). Proportions of specimens with squamocolumnar cells will be compared for the 5 cm and 3 cm swabs.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 23 | 27
Participants
  Presence of squamocolumnar cells - Yes | 11 | 8
  Presence of squamocolumnar cells - No | 12 | 19

2. Secondary Outcome: Cytologic Adequacy
Description: The presence of ~2000-3000 nucleated squamous cells will be assessed for cytologic adequacy (Yes/No). Proportions of adequate specimens will be compared for the 5 cm and 3 cm swabs.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 23 | 27
Participants
  Cytologic adequacy - Yes | 20 | 19
  Cytologic adequacy - No | 3 | 8

3. Secondary Outcome: User Acceptability of New NF Swab Compared to Swab From Prior Research
Description: Each participant will receive a short cytology CASI immediately after the cytology screening to rate their acceptability of the cytology screening on a Likert scale. Proportions of individuals' ratings for acceptability will be compared for the new NF swab vs the swab from the prior research.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 23 | 27
Participants
  Willing to do anal self-swabbing in the future - Strongly agree | 13 | 21
  Willing to do anal self-swabbing in the future - Agree | 10 | 6
  Willing to do anal self-swabbing in the future - Disagree | 0 | 0
  Willing to do anal self-swabbing in the future - Strongly Disagree | 0 | 0
  Willing to do anal self-swabbing in the future - Don't know | 0 | 0
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Equivalence — Equivalence is established if p>0.05; p = 0.99, Fisher Exact

4. Secondary Outcome: User Pain of New NF Swab Compared to Swab From Prior Research
Description: Each participant will receive a short cytology CASI immediately after the cytology screening to rate their pain during the cytology screening on a visual scale. Proportions of individuals' ratings for pain will be compared for the new NF swab vs the swab from the prior research.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 23 | 27
Participants
  No pain | 12 | 15
  A little pain | 9 | 10
  A little more pain | 1 | 1
  Even more pain | 1 | 1
  A whole lot of pain | 0 | 0
  Worst pain | 0 | 0
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Equivalence — Equivalence is established if p>0.05; p = 0.47, Chi-squared — Pain was dichotomized into a binary variable (0=no pain, 1=any amount of pain)

5. Secondary Outcome: User Pain by Swab Length
Description: Each participant will receive a short cytology CASI immediately after the cytology screening to rate their pain during the cytology screening on a visual scale. Proportions of individuals' ratings for pain will be compared for the 5 cm and 3 cm swabs.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 23 | 27
Participants
  No pain | 12 | 15
  A little pain | 9 | 10
  A little more pain | 1 | 1
  Even more pain | 1 | 1
  A whole lot of pain | 0 | 0
  Worst pain | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until 30 days after the intervention.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 0/23 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT07085845/Prot_SAP_000.pdf